CLINICAL TRIAL: NCT04233710
Title: Robotic Rehabilitation and Brain Stimulation for Children With Hemiparetic Cerebral Palsy
Acronym: RoboCP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Sean Dukelow, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REB17-1008
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Hemiplegic Cerebral Palsy; Perinatal Stroke
Keywords: robotic rehabilitation; tDCS; non-invasive brain stimulation
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot + tDCS (Experimental): 10 sessions of 1.5 hrs of robotic therapy within a 3 week period, with 20 minutes of 1mA cathodal tDCS applied to the contralesional M1 area during first 20 minutes of robotic therapy. Robotic therapy will be conducted using the Kinarm Exoskeleton robot and use games to target unilateral and bilateral motor and sensory impairments.
  Interventions: Combination Product: Robot Rehabilitation + tDCS
- Robot + sham tDCS (Sham Comparator): 10 sessions of 1.5 hrs of robotic therapy within a 3 week period with 20 minutes of SHAM tDCS applied during the first 20 minutes of the robotic therapy. As with experimental arm, electrode will be placed on contralesional M1. Current will ramp up and then immediately ramp down to simulate the cutaneous sensations felt with actual tDCS. Robotic therapy will be delivered with Kinarm Exoskeleton robot and use games to target unilateral and bilateral motor and sensory impairments.
  Interventions: Behavioral: Robotic Rehabilitation + sham tDCS

INTERVENTIONS:
Combination Product: Robot Rehabilitation + tDCS — Robotic therapy with Kinarm Exoskeleton Robot and 1 mA cathodal tDCS applied to contralesional M1 for 20 minutes.
  Arms: Robot + tDCS
Behavioral: Robotic Rehabilitation + sham tDCS — Robotic therapy with Kinarm Exoskeleton Robot and sham tDCS.
  Arms: Robot + sham tDCS

SUMMARY:
This study evaluates the use of robotic rehabilitation with and without transcranial direct current stimulation (tDCS) to improve motor performance in children with hemiparetic cerebral palsy. Half of the participants will receive robotic rehabilitation and half will receive robotic rehabilitation with tDCS. We hypothesize that tDCS may augment the robotic therapy and show greater improvements than robotic therapy alone.

DETAILED DESCRIPTION:
The defining feature of hemiparetic cerebral palsy is motor impairments primarily on one side of the body. Robotic rehabilitation and non-invasive brain stimulation are both emerging technologies that may be beneficial in improving motor performance in individuals with hemiparetic cerebral palsy. Robotic rehabilitation can allow for hundreds of arm movements in the span of an hour, a level of concentrated repetitions that is not possible in traditional rehabilitation. Additionally, robotics can target specific deficits, such as coordinating both arms together, improving accuracy of reaching movements, or improving proprioception, while simultaneously giving the therapist and patient quantitative feedback on performance. Non-invasive brain stimulation using transcranial direct current stimulation (tDCS) can safely modulate activity in regions of the brain and has emerged as a tool to enhance motor learning in typically developing children and augment therapy in children with hemiparetic cerebral palsy.

Children with hemiparetic cerebral palsy will be randomized to receive robotic rehabilitation with tDCS or robotic rehabilitation with sham-tDCS. Participants and the assessors will be blinded to the treatment. All children will complete 10 sessions within 3 weeks of 1.5 hours of robotic rehabilitation. The Kinarm Exoskeleton Robot will be used and children will play games with their affected arm or both arms to target different aspects of sensorimotor control. Children will simultaneously receive real or sham tDCS for the first 20 minutes of the session. tDCS will consist of 1 mA current with the cathode applied over the contralesional M1 area. All children will be assessed before and after the 10 session intervention period using robotic and clinical measures of motor and sensory performance, and at a 3 month follow up.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of hemiparetic cerebral palsy due to unilateral perinatal stroke
* age 6-18 years
* Manual Ability Classification System (MACS) Level I-III
* Modified Ashworth Score in shoulder and elbow <=3;
* Visual acuity (corrected) better than 20/50 in both eyes
* able to follow instructions and comply with protocol;
* able to give consent/assent;
* able to commit to all assessment and intervention sessions.

Exclusion Criteria:

* significant contractures in the upper extremity;
* other neurological conditions or active medical disease;
* unstable epilepsy;
* contraindications to tDCS;
* botulinum toxin A injections in the upper extremity in the past 6 months;
* upper extremity surgical intervention in past 6 months;
* involvement in another interventional study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Reaching Accuracy | change between pre-assessment (within 1 week of starting intervention) and post-assessment (within 1 week of completing intervention)
  Change in reaching accuracy as measured by initial direction error on robotic visually guided reaching task.

SECONDARY OUTCOMES:
Standardized robotic measures of motor and sensory performance | change between pre-assessment (within 1 week of starting intervention) and post-assessment (within 1 week of completing intervention)
  Robotic measures of spatiotemporal reaching (path length ratio, reaction time, movement speed, number of speed maximums), proprioception (variability in position matching) and bilateral object hitting task (number of balls hit with each hand). Each measure will be assessed as change from pre-assessment to immediate post-assessment
Assisting Hand Assessment | change between pre-assessment (within 1 week of starting intervention) and post-assessment (within 1 week of completing intervention)
  Performance on clinical assessment that determines how effectively the affected limb is used on tasks typically requiring both arms.
Box and Block Assessment | change between pre-assessment (within 1 week of starting intervention) and post-assessment (within 1 week of completing intervention)
  Measure of ability to reach, grasp and release that measures how many 1" cubes a child can move from one side of a box to another in 1 minute.
Purdue Pegboard | change between pre-assessment (within 1 week of starting intervention) and post-assessment (within 1 week of completing intervention)
  Measure of manual dexterity measured by how many small pegs a child can place in a pegboard in 30 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Dukelow, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Raess L, Hawe RL, Metzler M, Zewdie E, Condliffe E, Dukelow SP, Kirton A. Robotic Rehabilitation and Transcranial Direct Current Stimulation in Children With Bilateral Cerebral Palsy. Front Rehabil Sci. 2022 Feb 25;3:843767. doi: 10.3389/fresc.2022.843767. eCollection 2022. PMID 36188922